CLINICAL TRIAL: NCT00003893
Title: Sequencing of Chemotherapy and Radiotherapy in Adjuvant Breast Cancer
Brief Title: Adjuvant Chemotherapy Plus Radiation Therapy in Treating Women With Early-Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067062; CRC-TU-BR3015; EU-99005
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-11

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Doxorubicin; Epirubicin; Fluorouracil; Methotrexate; Mitomycin; Mitoxantrone; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Drug: mitomycin C
Drug: mitoxantrone hydrochloride
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumors cells. Combining chemotherapy with radiation therapy may kill more tumor cells. It is not yet known which regimen of chemotherapy plus radiation therapy is more effective for early-stage breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of adjuvant chemotherapy plus radiation therapy in treating women who have early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of synchronous vs sequential adjuvant chemotherapy and radiotherapy on local recurrence, disease-free and overall survival, and treatment delay in women with early-stage breast cancer.
* Compare the safety of these regimens, in terms of dose intensity and toxicity, in this patient population.
* Compare the quality of life and cosmetic outcome in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to clinical oncologist, axillary clearance (yes vs no), radiotherapy boost intent (boost vs no boost), and chemotherapy intent (cyclophosphamide, methotrexate, and fluorouracil [5-FU] vs anthracycline-containing regimen). Patients are randomized to one of two treatment arms.

Patients receive any chemotherapy regimen that includes cyclophosphamide, methotrexate, and 5-FU. Some regimens may also include epirubicin, doxorubicin, mitoxantrone, and/or mitomycin. Chemotherapy repeats every 3 weeks for 4-8 courses.

* Arm I (synchronous chemoradiotherapy): Patients receiving synchronous therapy receive any of the above chemotherapy regimens plus daily radiotherapy between courses 2 and 3 OR courses 5 and 6 of chemotherapy. Radiotherapy is administered for 3-5 weeks.
* Arm II (sequential chemoradiotherapy): Patients receiving sequential therapy receive any of the above chemotherapy regimens followed by daily radiotherapy beginning after completion of all chemotherapy (after course 6 or 8). Radiotherapy is administered for 3-5 weeks.

Treatment in both arms continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before chemotherapy, 2-3 weeks after the completion of all treatment, and then at 1, 2, and 5 years.

Patients are followed annually for 10 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 2,250 patients (1,125 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Early-stage disease

    * No metastatic disease
  * Complete surgical excision of tumor
* Planned use of adjuvant chemotherapy and radiotherapy
* If participating in the cosmetic outcome evaluation portion of the study, must have unilateral disease
* Hormone receptor status

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Bone marrow function adequate

Hepatic:

* Hepatic function adequate

Renal:

* Renal function adequate

Cardiovascular:

* Cardiac function adequate

Other:

* No other prior malignancy except basal cell or squamous cell skin cancer or carcinoma in situ
* No other medical or social condition that would preclude study compliance
* Fit to receive both adjuvant chemotherapy and radiotherapy (administered either synchronously or sequentially)
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy
* No concurrent epirubicin and doxorubicin as a study combination chemotherapy regimen

Endocrine therapy:

* Prior or concurrent hormonal therapy allowed
* No concurrent tamoxifen if treated with methotrexate, mitomycin, and mitoxantrone as a study combination chemotherapy regimen

Radiotherapy:

* See Disease Characteristics
* No concurrent internal mammary chain irradiation
* No concurrent orthovoltage irradiation to the whole breast

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* Concurrent participation in another clinical trial allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 1998-07; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indy Fernando, MD, Study Chair — University Hospital Birmingham
Locations (1):
- Queen Elizabeth Hospital at University of Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Background] Bowden SJ, Fernando IN, Burton A. Delaying radiotherapy for the delivery of adjuvant chemotherapy in the combined modality treatment of early breast cancer: is it disadvantageous and could combined treatment be the answer? Clin Oncol (R Coll Radiol). 2006 Apr;18(3):247-56. doi: 10.1016/j.clon.2005.11.010. PMID 16605056
- [Background] Fernando I, Bowden S, Dunn J: The combination of chemotherapy and radiotherapy in the adjuvant treatment of breast cancer. [Abstract] Radiother Oncol 58 (Suppl 1): A-34, S10, 2001.
- [Background] Fernando IN. The role of radiotherapy in patients undergoing mastectomy for carcinoma of the breast. Clin Oncol (R Coll Radiol). 2000;12(3):158-65. doi: 10.1053/clon.2000.9143. PMID 10942332
- [Derived] Fernando IN, Lax S, Bowden SJ, Ahmed I, Steven JH, Churn M, Brunt AM, Agrawal RK, Canney P, Stevens A, Rea DW. Detailed Sub-study Analysis of the SECRAB Trial: Quality of Life, Cosmesis and Chemotherapy Dose Intensity. Clin Oncol (R Coll Radiol). 2023 Jun;35(6):397-407. doi: 10.1016/j.clon.2023.03.007. Epub 2023 Mar 20. PMID 37012180
- [Derived] Fernando IN, Bowden SJ, Herring K, Brookes CL, Ahmed I, Marshall A, Grieve R, Churn M, Spooner D, Latief TN, Agrawal RK, Brunt AM, Stevens A, Goodman A, Canney P, Bishop J, Ritchie D, Dunn J, Poole CJ, Rea DW; SECRAB Investigators. Synchronous versus sequential chemo-radiotherapy in patients with early stage breast cancer (SECRAB): A randomised, phase III, trial. Radiother Oncol. 2020 Jan;142:52-61. doi: 10.1016/j.radonc.2019.10.014. Epub 2019 Nov 27. PMID 31785830